CLINICAL TRIAL: NCT03031873
Title: Evaluation of Susceptibility-weighted Magnetic Resonance Imaging and 4d-time-resolved Magnetic Resonance Angiography in Brain Arteriovenous Malformations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3T MRI evaluation
Record Dates: First submitted 2016-12-06; First posted 2017-01-26 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Arteriovenous Malformations
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI perfusion imaging (Other): SWAN imaging on the GE 3 T has been attempted but the preliminary evidence suggest that the images are of low resolution and difficult to interpret. Similarly, early experience with TRMRA suggest poor spatial and temporal resolution using the standard "out-of-the-box" protocols.
  Thus, there is a significant opportunity to improve SWAN and TRMRA, to evaluate the evolution of progressive obliteration of the AVM nidus. Specifically, this is attractive for brain AVMs that are treated with radiosurgery as MRI is required for clinical grounds for treatment planning purposes.
  Interventions: Device: MRI perfusion imaging

INTERVENTIONS:
Device: MRI perfusion imaging — Evaluate the evolution of progressive obliteration of the AVM nidus

SUMMARY:
Brain arteriovenous malformations are abnormal communications between brain arteries and veins with an intervening tangle of abnormal arteries (nidus). Brain AVMs may be asymptomatic or symptomatic, presenting with acute hemorrhage or neurological symptoms. Brain AVMs that have not bled carry a yearly risk of intracranial hemorrhage of approximately 4% (Ondra et al.).

The management is multidisciplinary involving neurosurgeons, interventional neuroradiologists, radiation physicians, neurologists and allied health care personnel. Patients may be treated with open neurosurgery, endovascular embolization, radiation therapy or any combination of these treatments. The goal of the treatment is to eliminate the brain AVM while preserving normal flow to the surrounding normal arteries. This involves obliteration of the shunting of blood via the AVM arteries to veins by a variety of treatments. The treatment regimen is individualized dependent on natural history, the angioarchitecture, location, risk of treatment(s) and patient wishes.

DETAILED DESCRIPTION:
Why is MRI important in the management of brain AVMs i.e. over conventional catheter angiography? The "gold standard" for evaluation of brain AVMs is catheter angiography. However, the procedure is invasive, involves ionizing radiation, exposure to contrast media with potential for nephrotoxicity or allergy and carries a 1% risk of morbidity including stroke. In contrast, MRI is a non-invasive method to evaluate brain AVMs and has the added advantage over catheter angiography of depicting the anatomical localization of the AVM within the brain tissue. However, currently MRI is limited by lack of ability to demonstrate shunting of blood through the AVM, an important indicator that the brain AVM is still present after treatment.

Susceptibility-weighted imaging (SWI) is a promising new MRI technology which indirectly evaluates the amount of oxygen within blood vessels. Small case series exploring the utility of SWI in brain AVMs has been reported suggesting the venous drainage of brain AVMs is often abnormally hyperintense because of abnormal shunting of oxygenated blood from AVM arteries to the draining vein(Bharathi D et al.). Typically in normal tissues, oxygenated blood on SWI images is hyperintense while deoxygenated blood in normal veins is hypointense. Developmental venous anomalies demonstrating enlarged draining veins are normal variants that must be distinguished from true AVMs . However, this capability has not been prospectively evaluated in a systematic fashion.

Our current standard for contrast-enhanced evaluation of brain AVMs is to perform a contrast-enhanced MRA (CEMRA) followed by a post-contrast T1 volumetric whole brain sequence. The CEMRA allows depiction of contrast at its maximal intensity passing through the brain on its first pass. The post contrast T1 scan only demonstrates static contrast pooling within the brain AVM. However, neither CEMRA nor the post contrast scan provides information about the speed at which contrast is moving through a brain AVM ie. shunting. Evaluation of the temporal passage of contrast brain AVM would require a dynamic time-resolved technique with adequate temporal resolution to distinguish early vs late vs no shunting within a brain AVM.

What is the current technology for MRI of brain AVMs? Susceptibility-weighted angiography (SWAN) imaging on the GE 3 T has been attempted but the preliminary evidence suggest that the images are of low resolution and difficult to interpret. In addition, our literature review found a paucity of studies evaluating staged treatment of brain AVMs with SWAN imaging. In our institution, brain AVMs may have staged treatment consistent of endovascular embolization and/or radiosurgery. After each treatment patients are followed with serial imaging MRI and Digital Subtraction Angiography (DSA). This provides an important opportunity to investigate the utility of non-invasive MRI to detect residual AVM after treatment.

Thus, there is a significant opportunity to evaluate the value of SWAN and Time Resolved Magnetic Resonance Angiography (TRMRA) assessment of progressive obliteration of the AVM nidus. Specifically, this is attractive for brain AVMs that are treated with radiosurgery as MRI and DSA are required for clinical grounds for treatment planning purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Brain AVMs previously diagnosed with either CT Angiography, MRI or catheter angiography.
3. Undergoing cerebral catheter angiography for clinical evaluation of the brain AVM. Patients with brain AVMs scheduled for catheter cerebral angiography will undergo MRI (GE 3T) within 3 months.
4. Age > 18 years.
5. mRS <=2
6. Brain AVM visible on MRI, i.e. nidus > 1 cm

Exclusion Criteria:

1. Contraindication to MRI eg. Non-MRI compatible implant, severe claustrophobia
2. Contraindication for contrast: GFR < 60 ml/min, allergy to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
SWAN and TRMRA with catheter angiography will be measured to determine if accuracy of brain MRI for follow-up of treated brain AVM can be improved | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lesiuk, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided